CLINICAL TRIAL: NCT06371508
Title: The Effect of Breast Cancer and Breast Self-examination Education Given to Women on Breast Cancer Fear and Breast Examination Skills
Brief Title: Breast Cancer and Breast Self-examination Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Yasemin Hamlaci Baskaya, Assist. Prof., Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14042024
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Breast Self-Examination
Keywords: breast self examination; breast cancer; education; fear
MeSH Terms: conditions — Breast Neoplasms; Breast Self-Examination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Women in the experimental group of the research will be given training content prepared by the researcher. The training presentation content will include information about breast cancer, breast cancer screening programs and breast self-examination.
  Interventions: Behavioral: Education based on breast cancer and breast examination
- Control group (No Intervention): Women in the control group will not be given any training and only their current information will be determined. Additionally, their awareness on this issue will be raised as they participate in the study.

INTERVENTIONS:
Behavioral: Education based on breast cancer and breast examination — Training for the intervention group will be provided with a 40-45 minute training organized by one of the researchers.
  Arms: Experimental group

SUMMARY:
According to a news published by the World Health Organization (WHO); More than 2.3 million cases of breast cancer occur each year, making it the most common cancer among adults. In 95% of all countries, breast cancer is the first or second cause of female cancer death. In 2020, 2.3 million women worldwide were diagnosed with breast cancer and 685,000 deaths occurred. In Turkey, breast cancer ranks first among the most common cancer types in women, and the number of breast cancer cases in women in 2020 was recorded as 74 638. As a result of this situation, WHO (2023) published the Global Breast Cancer Initiative Framework to save 2.5 million lives from breast cancer by 2040. This published framework includes health promotion for early detection, timely diagnosis and comprehensive management of breast cancer.

One of the most effective ways to reduce breast cancer mortality and morbidity rate is early diagnosis. It is important to determine early diagnosis and signs and symptoms of cancer before they appear. Early diagnosis of breast cancer is possible with breast self-examination (BSE), clinical breast examination and mammography. Breast self-examination is an important examination method in terms of detecting changes in breast tissue and preventing subsequent complications. It is also an easy-to-apply, cheap and non-invasive method. In Turkey, it is recommended that women regularly perform breast self-examination every month after the age of 20, women between the ages of 20 and 40 should have a clinical breast examination every two years, and women between the ages of 40 and 69 should have a clinical breast examination every year and have a mammogram every two years.

There are studies showing that fear of breast cancer has a positive and negative impact on early diagnosis behaviors. Champion et al. (2004) stated that women with moderate breast cancer fear had a high rate of early detection behavior, whereas low and high fear levels had a negative effect on behavior. In the study conducted by Yavan et al. (2010) on 188 women, 2% of the women. They found that 3 of them had regular BSE and 78.7% of them had never had a mammography. In addition, 85% of the women included in the study stated that they had a fear of breast cancer due to a family history of breast cancer, being diagnosed with breast cancer, and the presence of risk factors. Study results show that fear of breast cancer affects screening results. Therefore, aim in the study is; To determine the effect of breast cancer and BSE training given to women on breast cancer fear and BSE skills.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write,
* Having no history of breast cancer,
* No communication barriers,
* Not pregnant or lactating,
* Those who are willing and agree to participate in the research.

Exclusion Criteria:

* Having a mental illness,
* Those who wish to withdraw from any part of the research.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Champion Breast Cancer Fear Scale Change | pre-intervention, 1 month after intervention
  Breast Cancer Fear Scale; Champion et al. The scale developed by (2004) is an 8-item, one-dimensional, five-point Likert type measurement tool. The measurement tool was adapted to Turkish culture by Seçginli (2012). The items in the scale are scored by the participants as "strongly disagree" 1 point, "disagree" 2 points, "undecided" 3 points, "agree" 4 points, "completely agree" 5 points. The lowest score from the scale is 8 and the highest score is 40. As the scores from the scale increase, the level of breast cancer fear increases. 8-15 points from the scale indicate "low level of fear", 16-23 points indicate "medium level fear", and 24-40 points indicate "high level fear".
Breast Self Examination Checklist Success Score | pre-intervention, 1 month after intervention
  Breast self-examination proficiency rating instrument-BSEPRI was developed by Robin Wood in 1994. In the study, the form will be used to evaluate women's ability to perform breast self-examination according to appropriate stages and their ability to detect breast masses. There are 10 statements in the form that include the stages of performing BSE. 10 points are given for each stage of the examination that is completed correctly, and 0 points are given for any stage that is incorrectly performed or not performed. Accordingly, a minimum of 0 and a maximum of 100 points are taken from the form. A BSE score of 90 or above indicates that the BSE was performed correctly, and a score of 80 or below indicates that the BSE was not performed correctly.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Hamlacı Başkaya, Phd., Study Director — Sakarya University
Locations (1):
- Kocadere Sağlık Evi, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No